CLINICAL TRIAL: NCT00896298
Title: Double-Blind, Placebo-Controlled Trial of Leptin Replacement Therapy in Patients With Lipodystrophy
Brief Title: Trial of Leptin Replacement Therapy in Patients With Lipodystrophy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Abhimanyu Garg, Chairman, Division Nutrition and Metabolic Diseases, Professor Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0502-294
Record Dates: First submitted 2009-05-08; First posted 2009-05-11 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Hypoleptinemia; Generalized Lipodystrophy; Partial Lipodystrophy; Insulin Resistance
Keywords: Lipodystrophy; Insulin secretory response
MeSH Terms: conditions — Lipodystrophy, Congenital Generalized; Lipodystrophy, Partial, Acquired; Insulin Resistance; Lipodystrophy | interventions — Leptin; recombinant methionyl human leptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Leptin (Active Comparator): Active Comparator for 4 months, then for 8 months.
  Interventions: Drug: Leptin
- 2 Sugar pill (Placebo Comparator): Placebo for 4 months, then active comparator for 8 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Leptin — Leptin injected subcutaneously twice a day, to be administered at 100% of the estimated replacement dose during the first month, which is a dosage of 0.03mg/kg for female children, 0.04mg/kg for adult females, and0.02 mg/kg for all males, and then at 200% subsequently, or placebo.
  Other Names: Recombinant-methionyl Human Leptin.; r-metHuLeptin
  Arms: 1 Leptin
Drug: Placebo — Sugar pill
  Arms: 2 Sugar pill

SUMMARY:
Lipodystrophies represent a therapeutic challenge with regards to insulin resistance, hypertriglyceridemia and fatty liver which often is coupled with significant adipose tissue loss. The purpose of the study is to examine the safety and efficacy of Leptin on subjects with lipodystrophy.

DETAILED DESCRIPTION:
The mechanism by which leptin improves glucose and lipid control is not clear. We will examine the possible mechanisms of leptin action by studying the effects of leptin administration on food intake, insulin resistance, insulin secretory response, hepatic and intramuscular triglyceride stores in a large sample of patients with lipodystrophy.

Hypothesis: Leptin replacement in patients with generalized and partial lipodystrophy and hypoleptinemia will be safe and efficacious in improving the metabolic abnormalities associated with insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* age > 6 years
* Partial and generalized lipodystrophy
* Serum leptin levels less than the 7th percentile of normal values reported by the 3rd National Health and Nutrition Examination survey (less than 7.0 ng/mL in females and less than 3/0 ng/mL in males)
* Presence of at least one of the following metabolic abnormalities:

  1. Type 2 Diabetes Mellitus
  2. Fasting serum insulin >20 uU/mL
  3. Fasting serum triglycerides > 300 mg/dL
  4. Previous participation in leptin trial (Amgen 991265, GCRC 660) - for Part B of the Study.

Exclusion Criteria:

* Known liver disease due to causes other than non-alcoholic steatohepatitis.
* Hematocrit of less than 30%.
* Current alcohol or substance abuse.
* Use of anorexigenic drugs, anabolic steroids, GH and thiazolidinediones
* Active tuberculosis
* Psychiatric disorder impeding competence or compliance
* Malignancies
* HIV infection
* Subjects who have a known hypersensitivity to E. Coli derived proteins
* Other condition, which in the opinion of the clinical investigators would impede completion of the study.

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abhimanyu Garg, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Leptin Therapy: Randomized to Leptin Therapy for 4 months.
- Placebo: Randomized to Placebo for 4 months.
Period: Overall Study
Arm/Group | Leptin Therapy | Placebo
Started | 13 | 12
Completed | 10 | 9
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Leptin Therapy: Participants were randomized to receive Leptin .
- Placebo: Participants were randomized to receive Placebo .
- Total: Total of all reporting groups
Arm/Group | Leptin Therapy | Placebo | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.2 (11.9) | 24.9 (13) | 26.1 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 3 | 3 | 6
Body weight [Mean (Standard Deviation); unit: kg] | 65.5 (17.5) | 57.7 (16.0) | 61.8 (16.9)
Fasting serum Triglycerides [Median (Full Range); unit: mg/dL] | 309.3 [69.3 to 1096.7] | 443.8 [104.7 to 3556.3] | 309.3 [69.3 to 3556.3]
Fasting serum Glucose [Mean (Standard Deviation); unit: mg/dL] | 157.0 (74.2) | 184.0 (87.2) | 170.0 (80.2)
HbA1c [Mean (Standard Deviation); unit: % of haemoglobin] | 8.1 (2.5) | 8.0 (2.5) | 8.0 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Fasting Serum Triglycerides
Time Frame: 4 months
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Leptin Therapy | Placebo
Number analyzed (Participants) | 10 | 9
mg/dL | 203 [100 to 457] | 304 [129 to 3875]
Statistical Analysis 1: Comparison: Leptin Therapy vs Placebo; Test type: Superiority; p = 0.2572, Mixed Models Analysis

2. Primary Outcome: HbA1c
Time Frame: 4 months
Measure: Median (Full Range); unit: % of haemoglobin
Arm/Group | Leptin Therapy | Placebo
Number analyzed (Participants) | 10 | 9
% of haemoglobin | 8.1 [5 to 12] | 7.6 [5.1 to 11.5]
Statistical Analysis 1: Comparison: Leptin Therapy vs Placebo; Test type: Superiority; p = 0.71, Mixed Models Analysis

3. Secondary Outcome: Fasting Serum Glucose
Time Frame: 4 months
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Leptin Therapy | Placebo
Number analyzed (Participants) | 10 | 9
mg/dL | 162 [77 to 310] | 165 [77 to 327]
Statistical Analysis 1: Comparison: Leptin Therapy vs Placebo; Test type: Superiority; p = 0.68, Mixed Models Analysis

4. Secondary Outcome: Body Weight
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Leptin Therapy | Placebo
Number analyzed (Participants) | 10 | 9
kg | 62.5 (17.5) | 56.3 (17.6)
Statistical Analysis 1: Comparison: Leptin Therapy vs Placebo; Test type: Superiority; p = 0.0256, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 4 month
Arm/Group | Leptin Therapy | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 2/13 | 4/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Leptin Therapy (N=13) | Placebo (N=12)
viral illness, sinusitis, backache (Infections and infestations) | 1 (1) | 0 (0)
Headaches (General disorders) | 1 (13) | 0 (0) — Nausea and cramps
Pneumonia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Pneumonia twice. Went To ER and took oral antibiotics
Tonsillectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Right Ankle Pain (Surgical and medical procedures) | 0 (0) | 1 (1)
Blurry Vision and Epigastric pain (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days